CLINICAL TRIAL: NCT06229249
Title: Effectiveness of Carpal Ligament Self-myofascial Stretching Over Conventional Physical Therapy on Reducing Pain and Improving Function in Patients With Stage i and ii Carpal Tunnel Syndrome - a Comparative Study
Brief Title: Effectiveness of Carpal Ligament Self-myofascial Stretching in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AWH/EC/01/2022
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Myo-fascial stretching; Pain; Function
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The participants in this group received carpal ligament self-myofascial stretching along with conventional physical therapy.
  Interventions: Other: Carpal ligament self-myofascial stretching
- Control group (Active Comparator): The participants in this group received conventional physical therapy.
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Carpal ligament self-myofascial stretching — Carpal ligament self-myofascial stretching is a technique that involves applying pressure and stretching to the carpal ligaments and surrounding myofascial tissues of the wrist and hand. The objective is to release tension, improve flexibility, and alleviate discomfort or pain in the wrist and hand area.
  Arms: Experimental group
Other: Conventional physical therapy — In this technique, ultrasound therapy, nerve gliding exercise, tendon gliding exercise, and wrist splinting were performed.
  Arms: Control group

SUMMARY:
Carpal tunnel syndrome (CTS), also known as median mononeuropathy, occurs when the median nerve is squeezed or compressed as it travels through the carpal tunnel at the wrist. It is common in the age group of 40-60 years. The main aim of the study was to compare the effectiveness of carpal ligament self-myofascial stretching over conventional physical therapy on reducing pain and improving function in patients with stage I and II CTS-thirty-six subjects with stage I and II (mild) CTS were recruited. Thirty-six subjects who fulfilled the inclusion criteria were randomly assigned to the experimental group and control group, with 18 patients in each group. The experimental group received carpal ligament self-myofascial stretching along with conventional physical therapy, while the control group received traditional physical therapy alone. The duration of the treatment was six weeks. The outcome measures used were the Boston Carpal Tunnel Questionnaire and the Visual Analogue Scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CTS between age group 30 - 60 years.
* Patients with stage I and II (mild) CTS, confirmed by nerve conduction study (EMG diagnosed by a medical professional).
* Patients who are able to read and understand English.

Exclusion Criteria:

* Presence of polyneuropathy.
* Consistent use of adaptive equipment, such as wheel chair or cane.
* Patients presenting with shoulder pathologies.
* Patients with other neurological or musculoskeletal conditions including Cervical radiculopathy, History of wrist and hand fractures, Upper extremity joint dislocations, Brachial plexus injuries, Cubital tunnel syndrome, Rheumatoid arthritis, De quervain's tenosynovitis, Cut injuries of hand.
* Patients who have underwent recent carpal tunnel release (within 1 year).

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Questionnaire | 6 weeks
  The Boston carpal tunnel syndrome is a disease-specific patient-filled questionnaire, which comprises of two scales, a symptom severity scale (SSS) and a functional status scale (FSS). The symptom severity scale has 11 questions scored from 1 point (mildest) to 5 points (most severe) and the functional status scale has eight questions scored from 1 point (no difficulty with activity) to 5 points (cannot perform the activity at all). The greater the score, the more severe the severity of the disease.
Visual Analogue Scale | 6 weeks.
  The visual analogue scale consists of a 10-cm line, with the left extremity representing (the absence of pain) and the right extremity indicating (great pain). The greater the score, the more severe will be the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, MPTh, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No